CLINICAL TRIAL: NCT03382860
Title: Estimation of Intracranial Pressure Using Non-invasive Fundus Videos
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Statumanu Icp ApS (Unknown)
Responsible Party: Principal Investigator, Frantz Rom Poulsen, Professor, PhD, MD, Odense University Hospital
Other Study IDs: S-20170038; 2012-58-0018 (Other: Datatilsynet, Region of Southern Denmark)
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Intracranial Pressure
Keywords: Intracranial Hypertension; Intracranial pressure monitoring; Non-invasive point-of-care device; Normal pressure hydrocephalus
MeSH Terms: conditions — Intracranial Hypertension; Hydrocephalus, Normal Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ventriculoperitoneal dysfunction: Patients with suspected ventriculo-peritoneal (VP) shunt dysfunction are admitted to the neurosurgical department for intracranial pressure monitoring for 24 hours. The patients are approached within this time frame.
  Interventions: Diagnostic Test: Fundus videos
- Normal Pressure Hydrocephalus (NPH): Patients with suspected NPH (triad of cognitive dysfunction, urine incontinence of urge type, abnormal gait) are admitted to the neurosurgical department for intracranial pressure monitoring for 24 hours. The following day an infusiontest is performed, where data is collected.
  Interventions: Diagnostic Test: Fundus videos

INTERVENTIONS:
Diagnostic Test: Fundus videos — Recordings of fundus videos

SUMMARY:
The purpose of this pilot study is to assess whether the intracranial pressure (ICP) can be detected by using a non-invasive retinal fundus scanner, recording the vessels of the eye entering from the optic disc. The artery's diameter (A) is measured and compared to the vein's diameter (V) thereby a ratio A/V can be calculated. This ratio is compared to the values obtained from conventional fiberoptic intraparenchymal, intraventricular ICP monitoring using external ventricular drain (EVD) or lumbar pressure monitoring.

Valid non-invasive techniques for objective measurements of the intracranial pressure do not exist at the given time now and this study could prove to help the development of monitoring patients ICP without surgical intervention.

DETAILED DESCRIPTION:
Intracranial pressure (ICP) is based on the simple principle of Monroe-Kellie Doctrine. Since the volume of the cranial cavity is constant and the brain, CSF and blood can only compensate for a certain change in volume, pressure will increase at a critical increase in volume. An increase in pressure caused by an increase in intracranial volume is distributed throughout the entire brain and spinal canal equally. The normal range of ICP varies with age. Normal values are less than 10-15 mmHg for adults and adolescents, 3-7 mmHg for younger children and 1.5-6 mmHg for newborns even sub-atmospheric ICP has been shown.

The threshold for intracranial hypertension varies in the literature, which is reflected in the clinical use. Generally, ICP above 20 mmHg is defined intracranial hypertension. ICP higher than 20-25 may require treatment, and continuous ICP above 40 mmHg indicates severe, lethal intracranial hypertension.

Some forms of measurements, e.g. 1. Intraparenchymal strain gauge or fiber optics or 2. Intraventricular ICP monitoring via external ventricular drain (EVD). EVD is considered golden standard, but in the daily clinic there is often no or limited difference between 1. and 2. The issue regarding invasive methods are the same as for any surgical procedure, e.g. bleeding and infection. Risk of bleeding is 2-10% for EVD and 2.5% for intraparenchymal monitors. The consequences of such a bleed can be severe and result in disability. EVD has a higher risk of infection (5-20%) compared to intraparenchymal monitors (0-0.1%).

Non-invasive methods such as transcranial doppler ultrasound pulsation index and optic nerve sheath diameter has been used in studies, which seemed promising, but has not yet been validated for routine clinical use. Also, in non-invasive methods there are significant inter observational variation.

Studies of the eye's fundus have shown a correlation between ICP and ratio between artery and vein diameter (A/V ratio, unpublished data) Currently, there are no published work that has considered the correlation between A/V ratio and ICP, however there is a study with a theoretical prediction of such a correlation (Babbs CF 2016. Weldon School of Biomedical Engineering Faculty Working Papers. Paper 1 http://docs.lib.purdue.edu/bmewp/1).

This study investigates the correlation between non-invasive fundus ICP estimation and intracranial pressure monitoring.

In practice, all conscious and able adults admitted to Odense University Hospital for intracranial pressure monitoring/measurements by either an EVD, intraparenchymal ICP monitor or lumbar spinal fluid pressure assessment are enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older with indication for intraparenchymal or intraventricular ICP monitoring
* Conscious and able
* Admission to the Department of Neurosurgery or Department of Neurology at Odense University Hospital

Exclusion Criteria:

* Disabled and unconscious
* No intraparenchymal or intraventricular ICP monitoring

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All conscious and able patients of 18 years and older admitted for intracranial pressure monitoring in the department of neurosurgery (Camino, Integra, Switzerland)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Absolute A/V ratio value to conventional intracranial pressure monitors | 2025
  Comparison of A/V ratio values from the fundus video analysis and conventional intraparenchymal intracranial pressure (ICP), intraventricular ICP monitoring or lumbar pressure monitoring.

SECONDARY OUTCOMES:
Change in A/V ratio value compared to increased intracranial pressure monitor during infusion test. | 2025
  Assessment of the use of the fundus videos in patients undergoing a lumbar infusion test for 20 minutes for assessment of normal intracranial pressure compared to a conventional intraparenchymal ICP monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Odense University Hospital, Odense C, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
We wish to share all data of individual intracranial pressure values and A/V ratio.

REFERENCES:
- [Result] Andersen MS, Pedersen CB, Poulsen FR. A new novel method for assessing intracranial pressure using non-invasive fundus images: a pilot study. Sci Rep. 2020 Aug 3;10(1):13062. doi: 10.1038/s41598-020-70084-0. PMID 32747697
- See also: Biomechanics of Retinal Venous Pulsations as Indicators of Intracranial Pressure — http://docs.lib.purdue.edu/bmewp/1